CLINICAL TRIAL: NCT03655093
Title: Validation of a Self-questionnaire in French on the Use of the Upper Limbs in Patients With Multiple Sclerosis
Acronym: MS-SEP
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3063; 2017-A00788-45 (Other: ID RCB)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Self-questionnaire; Measurement tools
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple sclerosis: Patients with MS according to the diagnostic criteria of 2010 Validation of AMSQ questionnaire
  Interventions: Other: Validation of AMSQ questionnaire

INTERVENTIONS:
Other: Validation of AMSQ questionnaire — Participation in the study will be proposed to any patient meeting the inclusion criteria and consulting a neurologist from the SEP reference center of the University Hospital of Rennes.
  The neurologist will explain the purpose of the study to the patient, give him the information form.
  Without opposition from the patient, the neurologist will give him the self-questionnaire. The patient will fill it during the consultation. In case of disability to the upper limbs making it impossible to fill the questionnaire by the patient, it will be filled by the neurologist or the patient's companion, according to the answers given by the patient.
  While the patient completes the questionnaire, a record of clinical information will be filled in by the neurologist.
  No additional act will be performed except the questionnaire, which result will not change the patient's management.

SUMMARY:
Multiple sclerosis (MS) is an inflammatory and demyelinating disease of the central nervous system that causes disability in young adults. This disability can take many forms depending on the neurological systems affected: disability walking, cognitive impairment or disability in the upper limbs. The development of validated measurement tools for these different disabilities is essential for the follow-up of patients in clinical routine and for the evaluation of new therapies.

DETAILED DESCRIPTION:
A specific self-questionnaire for patients with MS has recently been developed and validated in English and Dutch: "The Arm Function in Multiple Sclerosis Questionnaire (AMSQ)". The questionnaire groups 31 items and was created from questionnaires developed for other pathologies. The Dutch team that developed this questionnaire combines biostatisticians and neurologists, experts in the development and validation of disability measurement tools.

This study aims to validate the French version of AMSQ questionnaire. This study is carried out in collaboration with the Amsterdam team, which has carried out the methodology and will conduct the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with MS according to the diagnostic criteria of 2010
* Age ≥18 years
* Patients seen in consultation at the SEP reference center in Rennes

Exclusion Criteria:

* Other neurological or rheumatological pathology hindering the use of the upper limbs
* Inability to understand
* Minors
* Major persons subject to legal protection (legal safeguards, guardianship)
* Persons deprived of their liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MS according to the diagnostic criteria of 2010
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-07-03 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Validate the French version of the AMSQ self-questionnaire in a population of MS patients | At inclusion
  Evaluate item fit of the French version of the AMSQ using the graded response model, developed by Samejima (cf. reference)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kerbrat, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Samejima F. Estimation of latent ability using a response pattern of graded scores. Richmond, VA: The Psychometric Society, 1969.